CLINICAL TRIAL: NCT04272879
Title: Home Oxygen Therapy - Home Mechanical Ventilation 2: A Phase 4 Study
Brief Title: HOT HMV 2: A Phase 4 Study
Acronym: HOT-HMV2
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 228411
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Group — Those requiring NIV following an acute exacerbation of COPD

SUMMARY:
Smoking related lung disease or Chronic Obstructive Pulmonary Disease (COPD) is characterised by periods of worsening symptoms termed exacerbations. In some patients these may be severe enough to require hospitalisation and support for their breathing. Patients who suffer a severe exacerbation requiring breathing support using mask ventilation (also termed non-invasive ventilation, NIV) have a high chance of being readmitted to hospital in the following 12 months. Recent evidence suggests that the provision of a breathing machine at home (home mechanical ventilation, HMV) may reduce the risk of readmission to hospital in selected patients.

Morbidity and mortality in the 12 months following a life-threatening exacerbation of COPD remain high. Recent data from the Lane Fox Clinical Respiratory Physiology Research Centre supports the addition of home non-invasive ventilation to standard care to improve admission-free survival in patients with persistent hypercapnia following a decompensated exacerbation of COPD.

The study is designed to evaluate the clinical implementation of the delivery of home non-invasive ventilation in COPD patients with persistent hypercapnia following an acute exacerbation of COPD to validate that the clinical benefit derived from the HOT-HMV trial is maintained when the home non-invasive ventilation is implemented into routine clinical practice.

DETAILED DESCRIPTION:
Following publication of the home oxygen therapy-home mechanical ventilation (HOT-HMV) trial, the purpose of this study is to evaluate the clinical service delivery of home non-invasive ventilation (NIV) therapy in patients who have recently undergone, and recovered, from a life-threatening exacerbation of COPD.

This prospective cohort observational study is designed to evaluate the clinical implementation of the delivery of home non-invasive ventilation in COPD patients with persistent hypercapnia following an acute exacerbation of COPD to validate that the clinical benefit demonstrated by the HOT-HMV trial is maintained when the home non-invasive ventilation is incorporated into routine clinical practice.

Patients who have an admission to hospital with an acute exacerbation of COPD requiring non-invasive ventilation will be referred for assessment. Eligible patients will be referred by the critical care or appropriate respiratory team to a monthly assessment clinic for assessment of chronic hypercapnia. The total UK sample size will be 200 participants. St Thomas' critical care unit managed between 80-100 patients per year with non-invasive ventilation for life threatening exacerbation of COPD. This study will run over 4 years; therefore it is anticipated that 200 patients will be enrolled into the trial over this period. Patients will also be referred from peripheral hospitals to the Lane Fox Unit as a regional centre for home ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspected or with proven diagnosis of COPD
* Admission to hospital with life-threatening exacerbation of COPD requiring acute NIV (at admission evidence of decompensated Chronic Respiratory Insufficiencies (PaCO2 > 6kPa, pH <7.35)
* Arterial partial pressure of carbon dioxide (PaCO2) > 6kPa at discharge from hospital
* Discharge from hospital without combined home non-invasive ventilation and home oxygen therapy
* Patient willing to consider home non-invasive ventilation in addition to home oxygen therapy
* Patient suitable for home oxygen therapy (appropriate risk assessment)

Exclusion Criteria:

* Patient already established on home non-invasive ventilation and home oxygen therapy
* Patient unable to support home non-invasive ventilation e.g. unable to apply mask, lacking social support
* Patient on palliative care pathway
* Patient outside of usual catchment area for Lane Fox Respiratory Service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an admission to hospital with an acute exacerbation of COPD requiring non-invasive ventilation will be referred for assessment. Eligible patients will be referred by the critical care or appropriate respiratory team to a monthly assessment clinic for assessment of chronic hypercapnia.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
12 month admission free survival | 12 months
  How many patients were not admitted to hospital during the 12 months following initiation of NIV and still alive

SECONDARY OUTCOMES:
Barriers to receiving HOT-HMV treatment | 12 months
  Evaluating what are the barriers for patients to receive HOT HMV treatment within a clinical service
What proportion of patients receive HOT-HMV as a proportion to those who received NIV acutely | 12 months
  Evaluating the proportion of patients who received NIV acutely vs those who are eligible to receive HOT HMV from the clinical service
What proportion of patients receive HOT-HMV as a proportion to those who are elgible to received HOT HMV | 12 months
  Evaluating the proportion of patients are eligble to receive HOT HMV vs those who actually receive HOT HMV from the clinical service
Cost of the clinical time and input to set patients up onto HOT HMV | 12 months
  What does it cost to set someone up onto HOT HMV
Length of clinical time taken to set patients up onto HOT HMV | 12 months
  How long does it take a clinician to set someone up onto HOT HMV
Report the clinical pathway and structure to deliver HOT HMV clinically | 12 months
  Establish a detail report outlining the clinical pathway and structure required of the clinical team to deliver HOT HMV clinically
Machine malfunction and failure | 12 months
  Determine the reliability of the NIV machines issued clinically by monitoring their malfunction and failure rates
Re admission to hospital | 28 days
  How many patients are readmitted to hospital within 28 days from set up onto HOT HMV
Tolerability of HOT HMV: How patients perceive they are tolerating the HOT HMV | 12 months
  How patients perceive they are tolerating the HOT HMV
Patients Quality of Life | 6 weeks, 3 months, 6 months and 12 months
  Patients health related QoL by completing the Severe Respiratory Insufficiency questionnaire (SRI)
Patients Quality of Life | 6 weeks, 3 months, 6 months and 12 months
  Patients health related QoL by completing the COPD assessment test (CAT).
Adherence to HOT HMV | 6 weeks, 3 months, 6 months and 12 months
  Patients Adherence to their HOT HMV prescription taken from the datacard in their machine

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, MD, Study Chair — Guys & St Thomas NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No